CLINICAL TRIAL: NCT06993103
Title: A Randomised Controlled Trial of Pasteurised Donor Human Milk as Supplementary Nutrition for Infants Born to Women With Diabetes in Pregnancy.
Brief Title: Pasteurised Donor Human Milk Supplementation for Term Babies
Acronym: PRESENT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Murdoch Childrens Research Institute (Other); La Trobe University (Other); University of Melbourne (Other); South Australian Health and Medical Research Institute (Other); Australian Red Cross Lifeblood (Unknown); Monash University (Other); The Royal Women Hospital (Unknown); Frances Perry House (Ramsay Health) (Unknown); Ramsay Hospital Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-607; 2024607 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2025-03-25; First posted 2025-05-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Hypoglycemia; Metabolic Complication; Cows Milk Allergy; Hospital Length of Stay; Neonatal Intensive Care Unit; Breastfeeding; Mental Health Issue
Keywords: Pasteurised donor human milk; Donor breastmilk
MeSH Terms: conditions — Milk Hypersensitivity; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized controlled intervention trial - control and intervention arm
Masking Description: This study has 2 treatment arms. In the intervention arm, pasteurised donor human milk (PDHM) is provided to infants needing nutritional supplementation for the first 5 days of life, compared to standard hospital care.
  Participants will not be blinded to study group allocation, because a key research question concerns the consumer experience of accessing PDHM, including how maternal behaviors differ when receiving PDHM. The idea is that having human milk is a "bridge" to exclusive breast milk feeding, rather than a path to continued formula feeding and shorter breastfeeding duration. Many outcomes, such as maternal mental health, breastfeeding impact of access to PDHM) cannot be assessed in a blinded study. The primary outcome is unlikely to be impacted by lack of clinician blinding.
  Outcome assessments (analysis of questionnaire responses, skin prick testing for cow's milk allergy) and statistical analyses will be done by assessors blinded to study group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDHM - Pasteurised donor human milk (Experimental): All infants in this group will get access to Pasteurised donor human milk (PDHM) as supplementary nutrition. PDHM will be made available to the intervention group from the time of randomisation until day 5 of life. Families will be provided with a sufficient supply of frozen PDHM for home use to ensure an exclusively human milk diet up to day 5 of life if their infant is discharged before day 5. Access to PDHM will cease after 120 hours of life, and the infant will be fed according to standard hospital protocols or as per parent's decision.
  Interventions: Dietary Supplement: Dietary Supplement: PDHM Pasteurised Donor Human Milk
- Standard Care (Active Comparator): All infants in this group will receive the standard care as per local unit policy, including supplemental nutrition (e.g. infant cow's milk formula or IV fluids) as recommended by the treating clinician
  Interventions: Other: Standard care Cow's milk based formula

INTERVENTIONS:
Other: Standard care Cow's milk based formula — Standard hospital care would be given as as per local unit policy at the site.
  Other Names: Standard Care_Formula milk
  Arms: Standard Care
Dietary Supplement: Dietary Supplement: PDHM Pasteurised Donor Human Milk — PDHM will be given to infants randomised to the intervention group
  Other Names: PDHM_Donor milk
  Arms: PDHM - Pasteurised donor human milk

SUMMARY:
PRESENT is a multi-center randomised controlled trial that aims to assess whether access to pasteurized donor human milk as supplementary nutrition in the first five days of life for term infants born to women with diabetes in pregnancy reduces the proportion of infants who are admitted to a neonatal unit for management of hypoglycemia compared with current standard hospital care. The trial will also assess other important outcomes including breastfeeding rates, maternal mental health, and infant cow's milk allergy.

There will be two treatment arms. In the intervention arm, PDHM will be made available to infants from randomisation until day 5 of life. Infants allocated to the control arm will receive care as per local unit policy, including supplemental nutrition as recommended by the treating clinician. After hospital discharge, participants will be asked to complete an electronic questionnaire at 2 & 6 weeks and 6 & 12 months after birth. Questionnaires will assess infant feeding practices, maternal quality of life [including anxiety and depression symptoms and health-related quality of life] along with infant cow's milk allergy symptoms.

DETAILED DESCRIPTION:
Diabetes in pregnancy is becoming increasingly common globally, with more than 40 000 infants born to women with gestational diabetes alone in Australia each year. These infants are at a high risk of hypoglycaemia and often require admission to the neonatal intensive care unit (NICU) and frequent blood tests for glucose monitoring. Many lack access to sufficient maternal milk partly due to delayed lactogenesis, leading to reliance on cow's milk formula, which may increase risks of cow's milk allergy, early breastfeeding cessation, and long-term metabolic complications.

Pasteurized Donor Human milk (PDHM) supplementation represents an alternative to infant formula when sufficient mother's own milk is not available. In Australia, donor milk is already in use for more vulnerable populations (those born very preterm or of a very low birth weight). However, PDHM is not currently available for term infants, despite strong clinician and community demand.

Expanding the availability of PDHM to term infants has the potential to improve health outcomes for a much larger proportion of the population, with potential benefits for mothers and infants including a reduction in admissions to neonatal intensive care units, a reduction in cow's milk allergy in infants, and improved maternal mental health and breastfeeding outcomes.

Our project will assess the provision of PDHM as in-hospital supplementation for term infants who would otherwise be given cow's milk formula. This trial will address a significant gap in neonatal care and provide evidence to determine whether broader PDHM use could improve both mothers' and infants' and long-term health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all the following criteria to be enrolled in this trial:

* Mother is >18 years at the time of consent
* Mother has diabetes in pregnancy (type 1, type 2 or gestational diabetes)
* Mother intends to breastfeed for at least 6 weeks at the time of consent.
* Infant is born at ≥ 37 weeks and weighs > 2.5kg
* Clinician caring for infant decides that supplementary nutrition (in addition to maternal breast milk) is required within the first 48 hours after birth.
* Parent/s provide/s a signed and dated informed consent form and has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

Mother/infant pairs meeting any of the following criteria will be excluded from the trial:

* Multiple pregnancy
* Mother has a condition that precludes maternal breast milk consumption e.g. HIV, receiving chemotherapy
* Infant has clinically significant congenital abnormality interfering with effective breastfeeding or breast milk consumption (e.g., cleft lip and palate, metabolic disorder) and/or requiring immediate care in a neonatal unit (e.g., congenital heart disease).
* Infant has received infant formula prior to randomisation.
* Infant admitted to neonatal intensive care prior to randomisation.
* More than 48 hours old at the time of recruitment

Ages: 0 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1444 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants admitted to neonatal unit for management of hypoglycaemia | From birth to 120 hours of life
  Proportion of infants in intervention and standard care groups admitted to a neonatal unit for management of hypoglycaemia.

SECONDARY OUTCOMES:
Duration of hypoglycaemia (<2.6 mmol/L) | From birth upto 120 hours of life
  Length of time until 3 consecutive total blood glucose >2.6 mmol/L (hours) from randomization
Proportion of infants requiring IV access for dextrose | From birth to 30 days after hospital discharge
  By assessing the proportion of infants cannulated for IV dextrose during hospital admission or re-admission within 30 days of discharge.
Episodes of phlebotomy | From birth up to 120 hours of life
  By assessing the number of episodes of phlebotomy during initial hospital admission to discharge (infant).
Hospital length of stay (infant) | From birth up to initial hospital discharge, up to 90 days of life
  Duration of hospital stay from birth to hospital discharge, measured in hours.
Hospital re-admission within 30 days | From birth to 30 days after discharge
  By assessing the proportion of infants with hospital re-admission within 30 days of discharge
Neonatal unit admission and length of stay (infant) | From birth to initial hospital discharge, up to 90 days of life
  By assessing the proportion of infants admitted to the neonatal unit. For those admitted: the duration of admission (hours) will also be recorded.
Breast milk feeding | Breast milk feeding at 120 hours of age (this means received any breast milk in previous 24 hours) and at 2 & 6 weeks and 6 months of age
  An electronic questionnaire/survey will ask about any breast milk and/or exclusive breast milk feeding on separate occasions, including -
  * Day of onset of secretory activation
  * Infant receiving breastmilk (any, exclusive) in the previous 24 hours
  * at 2 weeks
  * at 6 weeks
  * at 6 months of age
  * Total duration of any breast milk feeding
  When relevant, would ask the reasons for stopping breastfeeding
Use of Formula feeding | Infant formula feeding at 120 hours of age (received any infant formula in previous 24 hours), and at 2 & 6 weeks and 6 &12 months of age
  Any formula use; exclusive use of formula:
  * in 24 hours prior to discharge
  * at 2 weeks
  * at 6 weeks
  * at 6 months of age The timing of the first formula use (to estimate the duration of end of exclusive human milk-only feeding) will also be recorded.
Maternal mental health in the post-partum period GAD-7 | At 6 weeks and 6 months post delivery
  Assessment of maternal anxiety and depression symptoms using the Generalized Anxiety Disorder 7 questionnaire, where scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Maternal mental health in the post-partum period using PHQ-9 survey | At 6 weeks and 6 months post delivery
  Assessment of maternal anxiety and depression symptoms using the Patient Health Questionnaire 9, where scores 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively.
Maternal & Infant Health-related quality of life using AQoL-4D | At 6 weeks and 6 months post delivery
  The Assessment of Quality of Life Measure AQoL-4D questionnaire will be used to capture mother's and infants quality of life.
Maternal & Infant Health-related quality of life using TANDI | At 6 weeks and 6 months post delivery
  The Toddler and Infant questionnaire will be used to capture infant health-related quality of life
Infant growth up to 12 months | At 4, 8 and 12 months of age
  Infant weight at hospital discharge, 4, 8 and 12 months of age (self-reported)
Maternal metabolic health | At pre-birth, 6 and 12 months post delivery
  Maternal weight (self-reported)
Maternal metabolic health | At 6-8 weeks after delivery
  By assessing maternal glucose tolerance test
Infant cow's milk allergy using Questionnaires | At 6 and 12 months
  Using an electronic survey asking about the symptoms related to cow's milk allergy
Infant cow's milk allergy using SPT | At 6 and 12 months
  More assessment will done using a skin prick test if required to confirm allergy status
Infant cow's milk allergy using OFC challenge | At 6 and 12 months
  Infants with a positive skin test will be further invited for an oral food challenge assessment, if required, to confirm allergy status
Infant antibiotic use in the first 12-months of life | At 6 weeks, 6 and 12 months
  By assessing the parent's reports on the use of antibiotics
Proportion of infants hospitalised with an infection in the first year of life | At 6 weeks, 6 and 12 months of age
  By assessing the parents' report for -
  * Antibiotic use in the first 12 months of life
  * Hospitalisation for infection in the first 12 months of life

OTHER OUTCOMES:
Exploratory outcomes: To explore the experience of supplementing using Pasteurised donor milk supplementation | At 6 week to 3 months
  To explore and understand the Stakeholder experience of PDHM (parents in both arms of trial; staff including midwives, lactation consultants, neonatologists, neonatal nurses, obstetricians, managers) using in depth parent interviews and non-participant interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Koplin, PhD, Principal Investigator — Child Health Research Centre, University Of Queensland
Locations (4):
- Australia (4):
  - Royal Brisbane and Womens Hospital (QLD), Brisbane, Queensland
  - Greenslope Hospital (QLD), Brisbane, Queensland
  - Frances Perry House (VIC), Melbourne, Victoria
  - Royal Womens Hospital (VIC), Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
All information collected during this study, including individual participant's personal health information, will be kept confidential and will not be shared with anyone outside the study unless required by law. Participants will not be named in any reports, publications, or presentations that may come from this study.

REFERENCES:
- [Background] Griffith RJ, Harding JE, McKinlay CJD, Wouldes TA, Harris DL, Alsweiler JM; CHYLD Study Team. Maternal glycemic control in diabetic pregnancies and neurodevelopmental outcomes in preschool aged children. A prospective cohort study. Early Hum Dev. 2019 Mar;130:101-108. doi: 10.1016/j.earlhumdev.2019.01.010. Epub 2019 Feb 1. No abstract available. PMID 30716594
- [Background] Shah R, Harding J, Brown J, McKinlay C. Neonatal Glycaemia and Neurodevelopmental Outcomes: A Systematic Review and Meta-Analysis. Neonatology. 2019;115(2):116-126. doi: 10.1159/000492859. Epub 2018 Nov 8. PMID 30408811
- [Background] Forster DA, Moorhead AM, Jacobs SE, Davis PG, Walker SP, McEgan KM, Opie GF, Donath SM, Gold L, McNamara C, Aylward A, East C, Ford R, Amir LH. Advising women with diabetes in pregnancy to express breastmilk in late pregnancy (Diabetes and Antenatal Milk Expressing [DAME]): a multicentre, unblinded, randomised controlled trial. Lancet. 2017 Jun 3;389(10085):2204-2213. doi: 10.1016/S0140-6736(17)31373-9. PMID 28589894
- [Background] Gertz B, DeFranco E. Predictors of breastfeeding non-initiation in the NICU. Matern Child Nutr. 2019 Jul;15(3):e12797. doi: 10.1111/mcn.12797. Epub 2019 Apr 2. PMID 30767426
- [Background] De Bortoli J, Amir LH. Is onset of lactation delayed in women with diabetes in pregnancy? A systematic review. Diabet Med. 2016 Jan;33(1):17-24. doi: 10.1111/dme.12846. Epub 2015 Aug 18. PMID 26113051
- [Background] Clifford V, Klein LD, Brown R, Sulfaro C, Hoad V, Gosbell IB, Pink J. Donor and recipient safety in human milk banking. J Paediatr Child Health. 2022 Sep;58(9):1629-1634. doi: 10.1111/jpc.16066. Epub 2022 Jul 2. PMID 35779010
- [Background] Clifford V, Klein LD, Sulfaro C, Karalis T, Hoad V, Gosbell I, Pink J. What are Optimal Bacteriological Screening Test Cut-Offs for Pasteurized Donor Human Milk Intended for Feeding Preterm Infants? J Hum Lact. 2021 Feb;37(1):43-51. doi: 10.1177/0890334420981013. Epub 2020 Dec 22. PMID 33351688
- [Background] Urashima M, Mezawa H, Okuyama M, Urashima T, Hirano D, Gocho N, Tachimoto H. Primary Prevention of Cow's Milk Sensitization and Food Allergy by Avoiding Supplementation With Cow's Milk Formula at Birth: A Randomized Clinical Trial. JAMA Pediatr. 2019 Dec 1;173(12):1137-1145. doi: 10.1001/jamapediatrics.2019.3544. PMID 31633778
- [Background] Halken S, Muraro A, de Silva D, Khaleva E, Angier E, Arasi S, Arshad H, Bahnson HT, Beyer K, Boyle R, du Toit G, Ebisawa M, Eigenmann P, Grimshaw K, Hoest A, Jones C, Lack G, Nadeau K, O'Mahony L, Szajewska H, Venter C, Verhasselt V, Wong GWK, Roberts G; European Academy of Allergy and Clinical Immunology Food Allergy and Anaphylaxis Guidelines Group. EAACI guideline: Preventing the development of food allergy in infants and young children (2020 update). Pediatr Allergy Immunol. 2021 Jul;32(5):843-858. doi: 10.1111/pai.13496. Epub 2021 Mar 29. PMID 33710678
- [Background] Titmuss A, Longmore DK, Barzi F, Barr ELM, Webster V, Wood A, Simmonds A, Brown ADH, Connors C, Boyle JA, Oats J, McIntyre HD, Shaw JE, Craig ME, Maple-Brown LJ; PANDORA Study Research Team. Association between hyperglycaemia in pregnancy and growth of offspring in early childhood: The PANDORA study. Pediatr Obes. 2022 Oct;17(10):e12932. doi: 10.1111/ijpo.12932. Epub 2022 May 29. PMID 35644889